CLINICAL TRIAL: NCT01121614
Title: A Pilot Study to Compare Collateral Damage and Vessel Sealing Ability of LOTUS Ultrasonic Shears, Ethicon Harmonic Scalpel™ and LigaSure™ on Human Mesenteric Blood Vessels
Brief Title: Mesenteric Vessel Sealing by Three Instruments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Plymouth NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 06/Q2103/139
Record Dates: First submitted 2010-05-07; First posted 2010-05-12 (Estimated); Last update posted 2012-07-09 (Estimated); Status verified 2012-07

CONDITIONS: Surgery
Keywords: Harmonic scalpel; ultrasonic scalpel; LOTUS; LigaSure; vessel sealing; burst pressure; collateral damage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- LOTUS (Experimental): LOTUS ultrasonic instrument
  Interventions: Device: LOTUS
- Ethicon Harmonic Scalpel (Experimental): Ultrasonic instrument
  Interventions: Device: Ethicon Harmonic Scalpel
- LigaSure (Experimental): Bipolar feedback vessel sealing device
  Interventions: Device: LigaSure bipolar vessel sealing device

INTERVENTIONS:
Device: LOTUS — Device used to seal blood vessel
  Arms: LOTUS
Device: Ethicon Harmonic Scalpel
  Arms: Ethicon Harmonic Scalpel
Device: LigaSure bipolar vessel sealing device
  Arms: LigaSure

SUMMARY:
Ultrasonic cutting-coagulation devices (UCCD) are surgical instruments which use ultrasonic energy to cut through and coagulate tissue. An Ethicon version (trademarked "Harmonic Scalpel" and "Ultracision") is used in a variety of surgical procedures. Its surgical performance has been directly compared with that of electrically powered diathermy instruments in animal and clinical trials. LOTUS is a company based in Ashburton, Devon, which has developed a UCCD that works in a slightly different way to the Harmonic Scalpel. There are also bipolar feedback diathermy instruments which use electrical energy to seal blood vessels, such as LigaSure. The aim of this project is to obtain data to design a fully powered trial to answer the research question: do LOTUS and Ethicon UCCDs and LigaSure bipolar device reliably seal and divide blood vessels? The investigators will also be examining the degree of collateral tissue damage caused by each instrument.

Hypotheses

* LOTUS UCCD, Ethicon Harmonic Scalpel and LigaSure are equivalent at sealing and dividing mesenteric blood vessels.
* LOTUS UCCD, Ethicon Harmonic Scalpel and LigaSure cause equal amount of collateral damage when sealing and dividing blood vessels.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing laparoscopic or open colorectal resection

Exclusion Criteria:

* Pregnant or lactating women
* Patients under eighteen years of age
* History of coagulation abnormality
* Inability to understand the nature of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-04; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Bursting pressure of sealed vessel | 1 day
  Designated instrument is used to seal and divide a blood vessel which has been dissected from large bowel mesentery. The pressure at which the seal leaks is measured using a pressure transducer, this is known as the "bursting pressure"

SECONDARY OUTCOMES:
Success/failure to seal vessel | 1 day
  Instrument is used to seal and divide a blood vessel, this outcome is to see whether the seal is complete
Depth of collateral damage | After histological fixation is complete; within one week
  Energy-based surgical instruments cause a certain amount of thermal damage to the surrounding tissue, to compare the 3 instruments this depth of damage will be measured histologically

CONTACTS AND LOCATIONS:
Locations (1):
- Derriford Hospital, Plymouth, Devon, United Kingdom

REFERENCES:
- [Derived] Noble EJ, Smart NJ, Challand C, Sleigh K, Oriolowo A, Hosie KB. Experimental comparison of mesenteric vessel sealing and thermal damage between one bipolar and two ultrasonic shears devices. Br J Surg. 2011 Jun;98(6):797-800. doi: 10.1002/bjs.7433. Epub 2011 Mar 25. PMID 21442611